CLINICAL TRIAL: NCT04146831
Title: Phase II Study of Sintilimab, a PD-1 Inhibitor, as Second-line Treatment in FH-deficient Renal Cell Carcinoma
Brief Title: Sintilimab in FH-deficient Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor, Doctor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI30820191025
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Renal Cell Carcinoma; FH-deficient; Sintilimab
Keywords: FH-deficient; Sintilimab; Second-line
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Sintilimab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab (Experimental): Sintilimab is administered in this arm.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: intravenous, 200mg, every 3 week. Course of treatment: Stop the treatment until clinical or radiographic progression occurs.

SUMMARY:
This is a single-arm phase II clinical trial to evaluate the initial efficacy and safety of Sintilimab, a PD-1 Inhibitor, as Second-line Treatment in FH-deficient Renal Cell Carcinoma.

DETAILED DESCRIPTION:
Fumarate hydratase-deficient renal cell carcinoma (FH-deficient RCC) is a rare subtype of RCC characterized by germline/somatic mutation of the fumarate hydratase (FH) gene, and is an extremely aggressive tumor, with a propensity to disseminate early even in the setting of a small primary tumor.

Loss-of-function mutation of FH results in the accumulation of fumarate, impairment of oxidative phosphorylation, alteration of the metabolic state, and stabilization of hypoxia-inducible factor (HIF)-1α, thus activating angiogenic and oxidative stress response pathways. Unlike the robust response of clear cell RCC (ccRCC) to antiangiogenic agents, blocking the antiangiogenic pathway does not lead to better outcomes in FH-deficient RCC. Anti-mTOR agents are also ineffective.

Although the National Comprehensive Cancer Network (NCCN) guideline recommends the combination of bevacizumab plus erlotinib or everolimus for metastatic FH-deficient RCC, high-level evidence for standardized systematic therapy remains scarce.

In the present study, the investigators plan to assess the efficacy and safety of immunotherapy with Sintilimab as second-line treatment in FH-deficient RCC, and to explore potential biomarkers related to the treatment efficacy by means of detection, including but not limited to the next-generation sequencing, flow cytometry, etc.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. histopathological evidence of FH-deficient renal cell carcinoma, which was confirmed by Sanger or next-generation sequencing after initial screening by IHC.
3. included patients must be diagnosed with metastatic renal cell carcinoma or have a TNM stage IV (according to 2009 TNM Classification). Patients must have received treatment of targeted agents or immunotherapy (including cytokine therapy) before enrollment.
4. ECOG score ≤2;
5. life expectancy ≥ 3 months;
6. sign informed consent, and be able to follow the visit and related procedures stipulated in the program;
7. agree to collect tumor tissue, blood and other specimens required by this study and apply them to relevant studies;
8. important organs and bone marrow functions meet the following requirements: absolute neutrophil count (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin (HGB) ≥9g/dL;Liver function: serum total bilirubin (TBIL) ≤1.5 times normal upper limit (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 times ULN, serum albumin (ALB) ≥ 2.8g /dL. Renal function: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥40 mL/min

Exclusion Criteria:

1. patients with other malignant tumors with different primary sites or histology from the tumor evaluated in this study within 2 years of personal history, except those with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or cervical carcinoma in situ under good control;
2. major surgery or severe trauma within 4 weeks before enrollment;
3. immunosuppressive drugs were used within 4 weeks prior to the first dose of study therapy, excluding local glucocorticoids, inhaled or otherwise, or systemic glucocorticoids at physiological doses (i.e., no more than 10mg/ d prednisone or equivalent doses of other glucocorticoids);
4. known or suspected active autoimmune diseases (congenital or acquired), such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. Patients with type 1 diabetes with good insulin control can also be enrolled.
5. known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
6. allergic to any component of monoclonal antibody;
7. suffering from other uncontrolled serious diseases, including but not limited to: A) severe infection in the active phase or clinically poorly controlled; B) HIV infection (HIV antibody positive); C) acute or chronic active hepatitis b (HBsAg positive and HBV DNA>1*103/ml) or acute or chronic active hepatitis c (HCV antibody positive and HCV RNA>15IU/ml); D) active tuberculosis, etc.;
8. class iii-iv congestive heart failure (New York heart association classification), poorly controlled and clinically significant arrhythmia;
9. uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg);
10. had any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, etc. within 6 months before the selected treatment;
11. diseases requiring the use of warfarin (coumarin) for anticoagulant treatment;
12. uncontrolled hypercalcemia (more than 1.5 mmol/L of calcium or calcium greater than 12 mg/dL or adjusted serum calcium greater than ULN), or symptomatic hypercalcemia requiring continued bisphosphate treatment;
13. accompanied by other malignant tumors (except those that have been cured, such as cervical carcinoma in situ, non-melanoma skin cancer, etc.);
14. other acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may result in increased risk associated with study participation or study drug administration, or interference with the interpretation of study results, and ineligibility to participate in the study as determined by the investigator;
15. pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate (6 month progression-free survival rate) | Up to 24 months
  Disease progression was defined as the time from first administration of Sintilimab to progression of disease (PD) or death, according to the Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months
  Complete response (CR) or partial response (PR) by Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST).
Duration of response (DOR) | Up to 24 months
  DOR is defined as the time from the date of first remission to the date of disease progression or death.
Progression-free survival (PFS) | Up to 24 months
  PFS is defined as the time from first administration of Sintilimab to the date of disease progression or death according to the Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST).
Overall survival (OS) | Up to 24 months
  OS is defined as the time from first administration of Sintilimab to the date of death according to the Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST).
Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index 19 (FKSI-19) | Up to 24 months
  FKSI-19 score change over time from baseline to disease progression. The scale of FKSI-19 is from 0 to 48, and higher scores indicate worse quality of life.
Functional Assessment of Cancer Therapy- Kidney Symptom Index- Disease related Symptoms (FKSI-DRS) | Up to 24 months
  FKSI-DRS score change over time from baseline to disease progression. The scale of FKSI-DRS is from 0-36, and higher scores indicate worse quality of life.
EuroQol five-dimension scale (EQ-5D) | Up to 24 months
  EQ-5D-5L score change over time from baseline to disease progression. The EQ-5D-5L is consisted of five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Higher scores indicate poorer health.
Visual analogue scale (VAS) | Up to 24 months
  VAS pain score change over time from baseline to disease progression. The scale of VAS is from 0-10, and higher scores indicate worse symptom of pain.
Frequency of treatment-related adverse events (AEs) | Up to 24 months
  Records were made according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

OTHER OUTCOMES:
Exploratory objectives | Up to 24 months
  To explore the correlations of genes detected by next-generation sequencing, MRI-based response patterns and biomarkers of peripheral blood with the efficacy of Sinitilimab.